CLINICAL TRIAL: NCT03287700
Title: Designing a Randomised Controlled Trial to Examine the Benefit of Bilateral Cochlear Implantation Compared With Unilateral Cochlear Implantation in Adults With Severe to Profound Deafness
Brief Title: Designing a Trial of Bilateral Cochlear Implantation in Adults
Acronym: FOUNDATION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Nottingham (Other); University of Liverpool (Other); University of Southampton (Other); University of East Anglia (Other); National Cochlear Implant Users Association, United Kingdom (Unknown)
Responsible Party: Sponsor
Other Study IDs: 16IH004; PB-PG-0815-20039 (Other Grant/Funding Number: National Institute for Health Research (UK))
Record Dates: First submitted 2017-09-12; First posted 2017-09-19 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-03

CONDITIONS: Hearing Loss, Bilateral; Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Bilateral; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Focus group participants: Adults who have received a cochlear implant on the National Health Service (NHS) at an auditory implant service in the United Kingdom (UK) OR Adults who have been referred to a UK auditory implant programme for assessment for cochlear implantation but who have not yet been implanted
  Interventions: Other: No intervention
- Online patient survey participants: Adults who have received a cochlear implant on the National Health Service (NHS) at an auditory implant service in the United Kingdom (UK)
  Interventions: Other: No intervention
- Online clinician survey participants: Clinicians who deliver the current care pathway for cochlear implantation at auditory implant programmes providing NHS services in the UK
  Interventions: Other: No intervention
- Trial design workshop participants: Clinicians who deliver the current care pathway for cochlear implantation at auditory implant programmes providing NHS services in the UK
  Interventions: Other: No intervention
- Manufacturer's forum participants: Representatives of manufacturers of cochlear implants who provide devices on the NHS
  Interventions: Other: No intervention
- Care pathway working group participants: Clinicians who deliver the current care pathway for cochlear implantation at auditory implant programmes providing NHS services in the UK
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be administered to any group in this observational study.

SUMMARY:
In the UK, cochlear implantation is the standard treatment for adults with 'severe-to-profound' deafness. This level of deafness means that without a cochlear implant they have difficulty understanding what people are saying even when they wear hearing aids. The NHS provides a cochlear implant for one ear even though these adults are deaf in both ears. Two cochlear implants could help them understand speech in noisy environments, know where to look to see who is talking, and avoid hazards outdoors.

The decision about who can receive cochlear implants and how many they can receive is based on guidance from the National Institute for Health and Care Excellence (NICE). NICE agreed that providing two cochlear implants can provide additional benefits over providing just one implant. However, they decided that there is not enough evidence to show that these additional benefits are worth the additional cost of providing the second implant. NICE recommended that a clinical trial should be conducted to gather this evidence.

This study will consult with patients to explore whether the trial would be acceptable to future implant recipients. The study will also work with clinicians to design a trial comparing bilateral and unilateral implantation in adults. These clinicians will also be surveyed to assess the acceptability of the trial. A group of clinicians that span the range of professions involved in delivering the care pathway will be invited to attend a trial design workshop to establish a consensus on acceptable trial design elements from a clinical perspective. Representatives from cochlear implant manufacturers will be consulted to determine possible strategies for securing industry support for a future trial. Those who run cochlear implantation services will be engaged in a working group to gather information on the current care pathway to inform future assessments of whether bilateral implantation could be cost-effective.

DETAILED DESCRIPTION:
The study design comprises focus groups, online surveys, a trial design workshop, a manufacturer's forum, and a care pathway working group.

Focus groups Two focus groups will be conducted to explore issues around the acceptability of the two-arm trial recommended by NICE. The recruitment strategy will target both individuals who have been referred for a cochlear implant but have yet to receive one and also existing users of a cochlear implant. The focus groups will explore issues such as acceptance of randomisation, how to minimise the burden associated with participating, potential barriers to participation, and how to communicate the purpose of the trial clearly and effectively to prospective participants.

Online surveys Online surveys, informed by the focus groups, will be used to capture the views of the wider population of patients and of clinicians who deliver cochlear implant services on the acceptability of the trial. Both surveys will use open and closed questions. The surveys will explore the acceptability of the trial.

Trial design workshop Following the focus groups and surveys, an all-day workshop will be conducted with clinicians who deliver the current care pathway for cochlear implantation. The workshop will comprise a focus group and a trial design session. The focus group will seek to identify pertinent issues with the trial design from the perspective of the clinicians. The group will then be tasked with reaching a consensus on a trial design that would be both acceptable to them and which is feasible to conduct.

Manufacturer's forum Major manufacturers who supply cochlear implants to the NHS will be invited to attend a manufacturer's forum near the end of the study. They will be presented with the results of the acceptability assessment. The forum will explore whether the manufacturers would consider supporting the trial.

Care pathway working group A working group of cochlear implant service coordinators will be established to examine the existing decision analytic model commissioned by NICE and to identify the aspects of the model that require updating. The group will identify those parameters for which relevant information may be available from their own service records and will be tasked to reach a consensus on individual values for each parameter that would generally represent service provision across the providers. The group will also define plausible ranges for each parameter which could be used in future sensitivity analyses of any decision-analytic model.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be 18 years or older at the time consent is obtained.
* Patients who participate in the focus groups and/or online survey must have received a cochlear implant on the NHS in the UK or must be currently being assessed for eligibility to receive a unilateral cochlear implantation by an NHS service provider.
* Clinicians who participate in the trial design workshop and/or the online survey must be employed by a provider of NHS cochlear implantation services in the UK and be a clinically-trained professional who delivers one or more aspects of the cochlear implantation care pathway.
* Representatives from manufacturers who attend the industry forum must be employed by a manufacturer of cochlear implants and hold a role that includes responsibility for developing, co-ordinating, or managing research activity sponsored and/or funded by the manufacturer.
* Clinicians who participate in the care pathway working group must be employed by a provider of NHS cochlear implantation services in the UK and have a head of service or co-ordinator role in their cochlear implant service or have been delegated responsibility to contribute on behalf of a head of service / co-ordinator.

Exclusion Criteria:

• None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with bilateral severe to profound hearing loss that is eligible for cochlear implantation in the United Kingdom following guidance from the National institute for Health and Care Excellence (NICE), who have either already been implanted or who are being assessed for eligibility to be implanted.
  Clinicians who deliver cochlear implantation services on the National Health Service in the UK.
  Representatives of manufacturers of cochlear implant systems who supply implants to the National Health Service in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-08-02 (Estimated); Study Completion 2019-08-02 (Estimated)

PRIMARY OUTCOMES:
Acceptability of trial among patients | Day 1 (Point at which the patient completes the online patient survey)
  Proportion of surveyed patients who consider the proposed trial comparing bilateral cochlear implantation to unilateral cochlear implantation to be acceptable

SECONDARY OUTCOMES:
Acceptability of trial among clinicians | Day 1 (Point at which the clinician completes the online patient survey)
  Proportion of surveyed clinicians who consider the proposed trial to be acceptable
Issues related to acceptability from patient perspective | Day 1 (On the day(s) the patient focus groups are conducted)
  Major themes related to acceptability from the perspectives of patients assessed using qualitative methods
Issues related to acceptability from clinician perspective | Day 1 (On the day the trial design workshop is conducted)
  Major themes related to acceptability from the perspectives of clinicians assessed using qualitative methods

CONTACTS AND LOCATIONS:
Overall Officials: Padraig T Kitterick, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Medicines for Children Clinical Trials Unit, Clinical Trials Research Centre, University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided